CLINICAL TRIAL: NCT00611091
Title: Improving Posthospital Medication Management of Older Adults Through Health IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Fallon Clinic (Industry); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jerry Gurwitz, Chief, Division of Geriatric Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12603; 1R18HS017203 (AHRQ)
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Adverse Outcomes Post-hospital Discharge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Intervention Group - (receive intervention) randomized at patient level - includes all health plan members, aged 65+, hospitalized at the study site hospital and discharged to an outpatient health plan clinic provider.
  Interventions: Other: Electronic delivery of enhanced discharge information to the ambulatory physician
- C (No Intervention): Control Group - (do not receive intervention) randomized at patient level - includes all health plan members, aged 65+, hospitalized at the study site hospital and discharged to an outpatient health plan clinic provider.

INTERVENTIONS:
Other: Electronic delivery of enhanced discharge information to the ambulatory physician — Follow-up appointment needs/plans
  Other Names: HIT
  Arms: I
Other: Electronic delivery of enhanced discharge information to the ambulatory physician — Laboratory follow-up needs
  Other Names: HIT
  Arms: I
Other: Electronic delivery of enhanced discharge information to the ambulatory physician — New medications
  Other Names: HIT
  Arms: I

SUMMARY:
The incidence of drug-induced injury is high in the ambulatory geriatric population and is increased for elders upon transition from the hospital to the ambulatory setting. In this application, we describe an effort to build on our extensive experience in medication safety and HIT-based medication management to respond to the AHRQ RFA entitled Ambulatory Safety and Quality Program: Improving Quality through Clinician Use of Health IT (RFA-HS-07-006). In this study, we propose to develop and evaluate the value of an enhanced, HIT-based transitional care intervention superimposed on the ambulatory electronic medical record (EMR) to improve the quality and safety of medication management, focusing particularly on the transition from the inpatient to the ambulatory setting for older adults with multiple comorbid conditions who are prescribed high risk medications. We propose a randomized controlled trial of a HIT-based transitional care intervention with enhanced medication and therapeutic monitoring alerts to improve the quality and safety of patient monitoring and medication management. We postulate that the efficient and coordinated delivery of actionable health information to the clinician via use of HIT in the ambulatory setting can improve medication safety for the growing geriatric population. The specific aims for this study are to evaluate, among a population of older adults discharged from the hospital, the impact of an enhanced discharge information system initiated upon transition to the ambulatory setting: (1) on the rate of follow-up by an outpatient provider within 14 days of hospital discharge; (2) on the prevalence of appropriate monitoring for selected high risk medications at 30 days from the time of hospital discharge; (3) on the incidence of adverse drug events (ADEs) 30 days after discharge; and (4) on the rate of emergency department visits and hospital readmission within 30 days of discharge. A secondary aim for this study is to determine costs directly related to the development and installation of the HIT-based transitional care intervention. This research allows for the examination of an integrated HIT intervention on the quality of follow-up, outpatient clinician workflow, occurrence of ADEs, and health care utilization to gain insights into the effective use of clinical alerts and coordinated delivery of actionable information to outpatient clinicians in the management of ambulatory elderly patients subsequent to hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years old, member of the study site health plan, hospitalized at the study site hospital, discharged to an outpatient provider at the study site health plan clinic

Exclusion Criteria:

* does not meet inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 5077 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
rate of follow-up to an outpatient provider within 14 days of hospital discharge. | 1 year 3 months
prevalence of appropriate monitoring for selected high risk medications at 30 days from the time of hospital discharge. | 1 year 3 months
incidence of adverse drug events (ADEs) 45 days after discharge. | 1 year 3 months
rate of hospital readmission and emergency department (ED) within 30 days of discharge. | 1 year 3 months

SECONDARY OUTCOMES:
assess whether a HIT-based transitional care intervention is more effective in subgroups of patients (by level of comorbidity, number of medications, and use of specific high risk medications) | 1 year 3 months
determine costs directly related to the development and installation of the HIT-based transitional care intervention. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jerry H Gurwitz, MD, Principal Investigator — Meyers Primary Care Institute/University of Massachusetts Medical School
Locations (1):
- St Vincent's Hospital, Worcester, Massachusetts, United States